Kingdom of Saudi Arabia Ministry of Education Umm Al-Qura University



المملكة العربية السعودية وزارة التعليم جامعة أم القرى

## **Consent to Participate**

Study title: Effectiveness of Digital Versus Hybrid Interventions in Promoting Nutrition Knowledge Among Adolescent Girls: A Randomized Trial.

| St | udy Ethical Approval Nun | nber: HAPO-02-I | K-012-2023-10-1787. | |
|---|---|---|---|---|
| Do | cument Date: September 1 | 2023 | | |
| Pa | rticipant ID | ••••• | | |
| Ple | ase indicate your agreen | nent with the fol | llowing statements | |
| 1. | I acknowledge that I have read and understood the research idea mentioned above. I have had the opportunity to think about it, ask questions, and receive satisfactory answers. | | | |
| 2. | I understand that the participation in this project is voluntary and not mandatory at all, and I have the right to withdraw at any time without providing reasons and without any consequences for myself or my child. | | | |
| 3. | I understand that my daughter's participation is voluntary and not mandatory at all, and she has the right to withdraw at any time without providing reasons and without any consequences for myself or my daughter. | | | |
| 4. | I would like to see the results of the research. | | | |
| 5. | I consent to my daughter participating in the research described above. | | | |
| 6. | My signature below indicates that I have understood the study information and have decided to allow my daughter to participate in the study. | | | |
| | Participant name | Date | Signature | |
| | Child name | Date | Signature (Guardian) | |
| | Researcher name | Date | Signature | |
| | المرفقات : | | التاريخ : | : |